CLINICAL TRIAL: NCT06288009
Title: Outcomes of Running Locking Suture vs Standard Running Suture in Surgical Wounds: a Randomized Evaluator-blinded Split-wound Comparative Effectiveness Trial
Brief Title: Outcomes of Running Locking Suture vs Standard Running Suture in Surgical Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2135389
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Scarring
Keywords: Running Locking Suture
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two blinded observers will record their scores independently using the POSAS instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Layered Closure with Running Locking Suture on Side A (Experimental): For all participants, one wound side half will be labeled as A and the other side as B. The bottom (subcutaneous) layer of the entire wound will receive the normal stitching. For the upper (cutaneous) layer, Side A will be closed with a running locking suture, and Side B will be closed with a standard running suture.
  Interventions: Procedure: Running locking suture; Procedure: Standard running suture
- Layered Closure with Running Locking Suture on Side B (Experimental): For all participants, one wound side half will be labeled as A and the other side as B. The bottom (subcutaneous) layer of the entire wound will receive the normal stitching. For the upper (cutaneous) layer, Side B will be closed with a running locking suture, and Side A will be closed with a standard running suture.
  Interventions: Procedure: Running locking suture; Procedure: Standard running suture

INTERVENTIONS:
Procedure: Running locking suture — In running locking sutures, the first anchoring knot is made at one end of the wound, and a loop of suture is left from the beginning of the throw. The needle is then passed through the loop of suture, locking the suture in place. This is repeated until reaching the end of the wound, where the suture material is then tied to the loop using an instrument tie for the final throw.
Procedure: Standard running suture — In standard running sutures, the first anchoring knot is made at one end of the wound, and all of the suture material is pulled through after completing the throw. This is repeated until reaching the end of the wound, where the suture material is then tied.

SUMMARY:
When patients have surgery on the head and face, stitches are the standard way to close the wound. Wounds always result in a scar, but doctors are always looking for ways to reduce scarring. Several studies have been done to test ways to close wounds that reduce scarring. The most commonly performed closure technique uses running sutures, where a single strand of suture is continued along the length of the wound with a series of uninterrupted stiches. However, alternative closure techniques exist such as the running locking suture, which can offer advantages such as improved tension and thus reduce post-operative complications with better aesthetic outcome. In this study, half the wound will be stitched with standard running sutures and the other half will be stitched with running locking sutures. This will allow us to see if the side with running locking sutures heals with less scarring.

DETAILED DESCRIPTION:
Following cutaneous surgical procedures, scar formation is inevitable. Reducing the degree of scar formation and achieving the best aesthetic outcome remains prominent within the dermatological literature.

Wound closure can be achieved by a variety of suturing techniques. After the dermis is closed using deep sutures, the epidermis is closed with a second layer of sutures for additional reinforcement. Approximating the epidermis is commonly performed with running sutures, where a single strand of suture is continued along the length of the wound with a series of uninterrupted stiches.

Running locking sutures are another technique that can achieve secondary layer closure of wounds. Like the running suture, the first anchoring knot is made at one end of the wound, but rather than pulling all of the suture material through after completing the throw, a loop of suture is left from the beginning of the throw, and the needle is then passed through the loop of suture, locking the suture in place. This is repeated until reaching the end of the wound, where the suture material is then tied to the loop using an instrument tie for the final throw. This technique may achieve better hemostasis by improving eversion and providing more equal tension across all loops of the running suture.

To our knowledge, the impact of scar cosmesis and rate of post-operative complications using a running locking suture technique in comparison to using standard running sutures for primary linear repair of surgical wounds has not been studied. This study seeks to determine the effectiveness of an alternative suturing technique for epidermal approximation by using individuals as their own controls in a split-scar model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the head or neck with predicted primary closure
* Willing to return for follow up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant Women
* Unable to understand written and oral English
* Wounds with predicted closure length less than 3cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Observer Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  The primary endpoint will be the score of two blinded reviewers independently using the POSAS assessment. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability, and surface area). All items are scored on a scale ranging from 1 ("like normal skin") to 10 ("worst scar imaginable"). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.

SECONDARY OUTCOMES:
Patient Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  This is the patient portion of the POSAS assessment, which will be independently recorded. The patient scale of the POSAS consists of six items (pain, itch, thickness, color, stiffness, and irregularity). All items are scored on a scale ranging from 1 ("as normal skin") to 10 ("yes, very different"). The sum of the six items results in a total score of the POSAS patient scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.
Width of Scar as measured using Trace-to-Tape Method | 3 months
  The trace-to-tape method is an objective measure for linear postoperative scars. The mean scar width will be determined using the trace-to-tape method. The surface area of the scar will be collected by tracing the scar with a water-based gel pen. While still wet, the gel residue will be lifted from the skin with clear packing tape and transferred on a sheet of paper.
Complications or Adverse Events from Treatment | 3 months
  For example, if one half of the scar has more associated erythema, as measured using the Trace-to-Tape method, then it will be recorded. Other complications from the treatment will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis - Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States

REFERENCES:
- [Background] Kantor J Kantor, Jonathan.
- [Background] Joshi AS, Janjanin S, Tanna N, Geist C, Lindsey WH. Does suture material and technique really matter? Lessons learned from 800 consecutive blepharoplasties. Laryngoscope. 2007 Jun;117(6):981-4. doi: 10.1097/MLG.0b013e31804f54bd. PMID 17545862
- [Background] MacDougal BA. Locking a continuous running suture. J Am Coll Surg. 1995 Dec;181(6):563-4. No abstract available. PMID 7582234
- [Background] Schlechter B, Guyuron B. A comparison of different suture techniques for microvascular anastomosis. Ann Plast Surg. 1994 Jul;33(1):28-31. doi: 10.1097/00000637-199407000-00006. PMID 7944193
- [Background] Wong NL. The running locked intradermal suture. A cosmetically elegant continuous suture for wounds under light tension. J Dermatol Surg Oncol. 1993 Jan;19(1):30-6. doi: 10.1111/j.1524-4725.1993.tb03326.x. PMID 8454786